CLINICAL TRIAL: NCT07407452
Title: A Prospective, Open-label, Multicenter Phase II Clinical Study of Iparomlimab and Tuvonralimab (QL1706) Combined With Standard Chemotherapy or Combined With Intraperitoneal Perfusion Chemotherapy and Olaparib as Neoadjuvant Therapy for Advanced Ovarian Cancer
Brief Title: Iparomlimab and Tuvonralimab (QL1706) Combined With Standard Chemotherapy or Combined With Intraperitoneal Perfusion Chemotherapy and Olaparib as Neoadjuvant Therapy for Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Xiaoxiang Chen, Department Director, Jiangsu Cancer Institute & Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2026-001
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancers
Keywords: ovarian cancer; ICIs; Neoadjuvant therapy; QL1706; olaparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin; Cisplatin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1：QL1706+paclitaxel +carboplatin /cisplatin (Experimental): Cohort 1: ECOG PS 0 or 1, all-comers population, regardless of BRCA or HRD test results. Treatment: iparomlimab and tuvonralimab (5 mg/kg, Q3W, D1) + paclitaxel (175 mg/m², Q3W, D1) + carboplatin (AUC 5-6, Q3W, D1)/cisplatin (75 mg/m², Q3W, D1). Planned enrollment: 30 patients.
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706)Injection; Drug: paclitaxel; Drug: carboplatin; Drug: Cisplatin
- Cohort 2：QL1706+olaparib+intraperitoneal perfusion (Experimental): Cohort 2: ECOG PS 2, BRCA1/2 mutation or HRD positive. Treatment: iparomlimab and tuvonralimab (5 mg/kg, Q3W, D1) + olaparib (300 mg, for 2-3 cycles, bid) + intraperitoneal perfusion (cisplatin, 75 mg/m², Q3W, D1). Planned enrollment: 20 patients.
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706)Injection; Drug: Olaparib; Drug: Cisplatin

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706)Injection — 5 mg/kg, Q3W, D1
  Other Names: QL1706
Drug: paclitaxel — 175 mg/m², Q3W, D1
  Arms: Cohort 1：QL1706+paclitaxel +carboplatin /cisplatin
Drug: carboplatin — AUC 5-6, Q3W, D1
  Arms: Cohort 1：QL1706+paclitaxel +carboplatin /cisplatin
Drug: Cisplatin — 75 mg/m², Q3W, D1
  Arms: Cohort 1：QL1706+paclitaxel +carboplatin /cisplatin
Drug: Olaparib — 300 mg, for 2-3 cycles, bid
  Arms: Cohort 2：QL1706+olaparib+intraperitoneal perfusion
Drug: Cisplatin — intraperitoneal perfusion, 75 mg/m², Q3W, D1
  Arms: Cohort 2：QL1706+olaparib+intraperitoneal perfusion

SUMMARY:
This study is a prospective, open-label, multicenter Phase II clinical trial, planning to enroll 50 patients with advanced ovarian cancer. Enrolled participants will be assigned to 2 cohorts based on ECOG performance status and genetic mutation status:

Cohort 1: ECOG PS 0 or 1, all-comers population, regardless of BRCA or HRD test results. Treatment: iparomlimab and tuvonralimab (5 mg/kg, Q3W, D1) + paclitaxel (175 mg/m², Q3W, D1) + carboplatin (AUC 5-6, Q3W, D1)/cisplatin (75 mg/m², Q3W, D1). Planned enrollment: 30 patients.

Cohort 2: ECOG PS 2, BRCA1/2 mutation or HRD positive. Treatment: iparomlimab and tuvonralimab (5 mg/kg, Q3W, D1) + olaparib (300 mg, for 2-3 cycles, bid) + intraperitoneal perfusion (cisplatin, 75 mg/m², Q3W, D1). Planned enrollment: 20 patients.

Neoadjuvant therapy will be administered for 3 cycles, followed by patient status assessment. Patients with CR/PR/SD will be allowed to undergo surgery, while PD patients will have subsequent treatment strategies determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily join this study, sign the informed consent form, and strictly comply with the protocol requirements;
* Female patients aged between 18 and 75 years;
* Patients who have undergone open surgery, laparoscopic surgery, or core needle aspiration biopsy, and have been histopathologically confirmed as having epithelial ovarian cancer (high-grade serous adenocarcinoma, endometrioid adenocarcinoma), peritoneal cancer, or fallopian tube cancer, FIGO 2018 Stage III-IV;
* Meet the indications for neoadjuvant chemotherapy in ovarian cancer: ① Preoperative assessment by gynecologic oncologists (with multidisciplinary consultation when necessary) indicates low likelihood of achieving R0 resection with primary debulking surgery; ② Physical condition unable to tolerate PDS, unsuitable for immediate surgery (e.g., high perioperative risk, advanced age, medical comorbidities, etc.); ③ No prior systemic anti-tumor treatment for ovarian cancer (including but not limited to radiotherapy, chemotherapy, surgery, targeted therapy, and immunotherapy); Note: Lymph node dissection or biopsy performed for clinical staging purposes after obtaining histopathology via needle biopsy, laparoscopic exploration, or other methods is permitted;
* Accept BRCA1/2 genetic mutation or HRD testing;
* Presence of at least one measurable lesion according to RECIST 1.1 criteria;
* Expected survival time ≥12 weeks;
* ECOG score 0-1 (for Cohort 1), ECOG score 2 (for Cohort 2);
* Adequate organ function, including:

Bone marrow function: Absolute neutrophil count ≥1,500/μL; Platelets ≥100,000/μL; Hemoglobin ≥10 g/dL Hepatic function: Total bilirubin ≤1.5× upper limit of normal (ULN) or direct bilirubin ≤1.0× ULN; AST and ALT ≤2.5× ULN; Must be ≤5× ULN when liver metastases are present Renal function: Serum creatinine ≤1.5× ULN, or creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula);

* Participants of childbearing potential must use appropriate contraceptive methods during the study period and for 120 days after study completion, have a negative serum pregnancy test within 7 days before study enrollment, and must be non-lactating participants.

Exclusion Criteria:

* Non-epithelial origin ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (e.g., germ cell tumors); ovarian tumors of low malignant potential (e.g., borderline tumors);
* Concurrent use of other cancer neoadjuvant therapies during this study, including but not limited to chemotherapy, radiotherapy, immunotherapy, microbial therapy, traditional Chinese medicine, and other experimental therapies;
* Hypersensitivity to the active or inactive ingredients of the investigational drug or drugs with similar structure to the investigational drug;
* Inability to swallow oral medications and any gastrointestinal disorders that may interfere with the absorption and metabolism of study drugs (for Cohort 2);
* Prior treatment with known or suspected poly (ADP-ribose) polymerase (PARP) inhibitors (for Cohort 2);
* Presence of symptomatic or uncontrolled brain metastases requiring concurrent treatment;
* Active or potentially recurrent autoimmune disease; exceptions include: vitiligo, alopecia, psoriasis, or eczema not requiring systemic treatment; hypothyroidism caused by autoimmune thyroiditis requiring only stable dose hormone replacement therapy; Type 1 diabetes requiring only stable dose insulin replacement therapy;
* Major surgery within 3 weeks before study initiation, or incomplete recovery from surgery;
* History of organ transplantation, autologous/allogeneic stem cell transplantation;
* Known or self-reported human immunodeficiency virus (HIV) infection;
* HBV-DNA positive, HCV-DNA positive (copy number >10³);
* Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40, etc.), immune cell therapy, or any other treatments targeting tumor immune mechanisms;
* Live vaccine administered within 4 weeks before first dose, or planned live vaccine administration during the study period;
* History of other malignancies within the past 3 years, except for cutaneous squamous cell carcinoma, basal cell carcinoma, ductal carcinoma in situ of the breast, or cervical carcinoma in situ;
* Prior or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
* Patients who received platelet or red blood cell transfusions within 4 weeks before initiation of study drug treatment;
* Pregnant, lactating, or patients planning to become pregnant during study treatment;
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | From enrollment to the end of treatment at 9 weeks
  Incidence and severity of AEs and TEAEs, vital signs, and clinically significant abnormal laboratory findings during the study period

SECONDARY OUTCOMES:
ORR | From enrollment to the end of treatment at 9 weeks
R0 Resection Rate | Periprocedural
DCR | From enrollment to the end of treatment at 9 weeks
12month-OS | From enrollment to the end of treatment at 12 month
24month-OS | From enrollment to the end of treatment at 24 month
OS | From enrollment to the end of treatment at 36 month
12month-PFS | From enrollment to the end of treatment at 12 month
PFS | From enrollment to the end of treatment at 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided